CLINICAL TRIAL: NCT01764867
Title: Algorithm Guided Treatment Strategies for Major Depressive Disorder
Acronym: AGTs-MDD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Yiru FANG, Ph.D., Professor of Psychiatry, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012BAI01B04-MDD; 2012BAI01B04 (Other Grant/Funding Number: 2012BAI01B04)
Record Dates: First submitted 2012-12-15; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Major Depressive Disorder
Keywords: major depressive disorder; algorithm guided treatment; treatment as usual; escitalopram; mirtazapine; transcranial magnetic stimulation (rTMS); modified electroconvulsive therapy (mECT); remission; relapse; quality of life
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Escitalopram; Mirtazapine; Transcranial Magnetic Stimulation; Fluoxetine; Citalopram; Paroxetine; Sertraline; Fluvoxamine; Venlafaxine Hydrochloride; Duloxetine Hydrochloride; Bupropion; Trazodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Algorithm Guided Treatment (AGT) (Active Comparator): Algorithm Guided Treatment (AGT) strategies include two steps. In the first step, participants will be randomly assigned to escitalopram (10-20mg/d) or mirtazapine (30-45mg/d) group. In the second step those non-remitted will be allocated into a set of different intervention groups including mirtazapine monotherapy (only for those taken escitalopram in the first step), escitalopram monotherapy (only for those taken mirtazapine in the first step), or combination therapies (i.e. escitalopram plus mirtazapine, escitalopram or mirtazapine plus either modified electroconvulsive therapy with 6-10 sessions or repetitive transcranial magnetic stimulation with 20 sessions respectively) according to intent-to-treat principle. Medication dosage in combination therapy has the same range as the first.
  Interventions: Drug: Escitalopram; Drug: Mirtazapine; Other: modified electroconvulsive therapy; Other: repetitive transcranial magnetic stimulation
- Treatment As Usual (TAU) (Active Comparator): This control arm refers to routine antidepressant treatment strategies for participants. Any of the new-generation antidepressants including fluoxetine, citalopram, escitalopram, paroxetine, sertraline, fluvoxamine, venlafaxine, duloxetine, mirtazapine, bupropion, or trazodone, which are all available in Chinese psychiatric clinics, may be used for participants who are randomly assigned to this treatment arm based on clinician's expertise and clinical judgement. The dosage range of any of the above antidepressants depends on clinician's judgement. The follow-up period will last up to 6-12 weeks. During follow-ups, clinician can decide to continue current treatment or start a switch or combination strategy based on his/her own clinical judgement.
  Interventions: Drug: Fluoxetine; Drug: Citalopram; Drug: Escitalopram; Drug: Paroxetine; Drug: Sertraline; Drug: Fluvoxamine; Drug: Venlafaxine; Drug: Duloxetine; Drug: Mirtazapine; Drug: Bupropion; Drug: Trazodone

INTERVENTIONS:
Drug: Escitalopram — Recommended dosage range of escitalopram is 10-20mg per day. The duration will last up to 6-12 weeks until progression or unacceptable intolerability develops.
  Other Names: Lexapro
  Arms: Algorithm Guided Treatment (AGT)
Drug: Mirtazapine — Recommended dosage range of mirtazapine is 30-45mg per day. The duration will last up to 6-12 weeks until progression or unacceptable intolerability develops.
  Other Names: Remeron
  Arms: Algorithm Guided Treatment (AGT)
Other: modified electroconvulsive therapy — Up to 6-10 sessions of mECT will be performed for selected participants who fails to remit to initial AGT intervention during 6 to 12-week period.
  Other Names: mECT
  Arms: Algorithm Guided Treatment (AGT)
Other: repetitive transcranial magnetic stimulation — Up to 20 sessions of rTMS will be performed for selected participants who fails to remit to initial AGT intervention during 6 to 12-week period.
  Other Names: rTMS
  Arms: Algorithm Guided Treatment (AGT)
Drug: Fluoxetine — Fluoxetine may be prescribed for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Citalopram — Citalopram may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Escitalopram — Escitalopram may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Paroxetine — Paroxetine may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Sertraline — Sertraline may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Fluvoxamine — Fluvoxamine may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Venlafaxine — Venlafaxine may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Duloxetine — Duloxetine may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Mirtazapine — Mirtazapine may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Bupropion — Bupropion may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)
Drug: Trazodone — Trazodone may be used for participants who are randomly assigned to the Treatment As Usual (TAU) arm based on clinician's judgement.
  Arms: Treatment As Usual (TAU)

SUMMARY:
The purpose of this study is to compare treatment outcomes between measurement based Algorithm Guided Treatment and Treatment As Usual strategies in a Chinese population with major depressive disorder.

DETAILED DESCRIPTION:
The AGT arm includes a 2-step medication monotherapy and a combination treatment algorithm. The first step (level 1) includes two medication monotherapy options: escitalopram and mirtazapine. For those participants who don't remit with the initial intervention after up to 6 to 12-week treatment, the second step (level 2) with a variety of treatment options will be provided. In level 2 intervention, a switch strategy for those who don't remit with escitalopram will be switched to mirtazapine, or for those who don't remit with mirtazapine will be switched to escitalopram, combination strategy (i.e. escitalopram plus mirtazapine) and augmentation strategy (i.e. escitalopram or mirtazapine plus either rTMS or mECT). Participants who don't get remission in level 1 intervention will be encouraged to enter level 2 interventions based on intend-to-treatment principle. The TAU arm as control intervention is performed using the psychiatrist's individual discretion based on his/her expertise and knowledge.

Participants will be recruited consecutively in 8 psychiatric settings across China and randomized into any of the two initial interventions of AGT or TAU arm. Follow-up interviews will be performed monthly for all participants who finish any acute treatment of AGT or TAU. The follow-up period will last up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for single or recurrent nonpsychotic major depressive disorder
* Age 18-75
* Written informed consent completed
* Scores 14 or higher on the 17-item Hamilton Depression Rating Scale
* Initial treatment with escitalopram or mirtazapine or other antidepressants is clinically appropriate

Exclusion Criteria:

* History of bipolar disorder
* Concurring psychotic disorders
* Scores 3 or higher on item 3 (suicidal) of HRSD-17
* History of nonresponse to an adequate trial of escitalopram and/or mirtazapine
* Has general medical condition, which contraindicates any leve 1 or 2 treatment option
* Is on concomitant medication, which contraindicates any leve 1 or 2 treatment option
* Any contraindication for mECT or rTMS
* Is pregnant or breast feeding or is planning to get pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Remission defined as endpoint 17-item Hamilton Rating Scale for Depression (HRSD-17) total score ≤ 7 | 12 weeks
  Acute treatment will last at least 6 weeks if remission occurs, or up to 12 weeks. Endpoint total score in HRSD-17 at up to 12 weeks will be measured to determine wether remission occurs.

SECONDARY OUTCOMES:
Remission defined as endpoint the Quick Inventory of Depressive Symptomatology (16-item) (QIDS-SR16) total score ≤ 5 | 12 weeks
Frequency and intensity of adverse events | 12 weeks
  Self-report and clinician rating frequency and intensity of adverse events will be measured at up to 12 weeks.
Quality of life | 12 weeks
  Change from baseline in 6-item Quality of life Inventory will be measured at up to 12 weeks.

OTHER OUTCOMES:
Relapse rate | 6 months
  Relapse rate will be measured at the end of 6 months after remission.

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, Ph.D., M.D., Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, China

REFERENCES:
- [Derived] Zhu Y, Wang F, Wang F, Liu H, Guo X, Wang Z, He R, Wu X, Cao L, Wu Z, Peng D, Fang Y. Program of algorithm for pharmacological treatment of major depressive disorder in China: Benefits or not? Heliyon. 2023 Oct 17;9(11):e20951. doi: 10.1016/j.heliyon.2023.e20951. eCollection 2023 Nov. PMID 37920522